CLINICAL TRIAL: NCT05364814
Title: The Effect of Using Probiotic Yogurt on Anthropometric Measurements and Gastrointestinal System in Obese Women
Brief Title: Use of Probiotic Yogurt in Obese Women
Status: Completed | Type: Observational
Sponsor: Yuksek Ihtisas University (Other)
Collaborators: Malatya Egitim Ve Arastirma Hastanesi (Other Government); Turgut Ozal University (Other)
Responsible Party: Principal Investigator, Sevan ÇETİN ÖZBEK, Assistant Proffesor, Yuksek Ihtisas University
Other Study IDs: YuksekIU02
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Dysbioses
MeSH Terms: conditions — Obesity; Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese Group: A single sample group . Anthropometric measurements were taken at the beginning of all patients. Yogurt with probiotic added to medical nutrition therapy was applied for 2 weeks.Anthropometric measurements were taken at the beginning of all patients. Yogurt with probiotic added to medical nutrition therapy was applied for 2 weeks. At the end of each week, food consumption records and scales were applied. During the wash out period, all patients were asked to comply with their diet only. After the wash out period, a different diet was started and the same procedures were repeated.During the wash out period, all patients were asked to comply with their diet only. After the wash out period, a different diet (with the addition of probiotic yogurt) was changed and the same procedures were repeated.

SUMMARY:
This study aimed to examine the effects of using probiotic yogurt on body components (body weight, height, etc.) and digestive system (distention, gas, etc.) in obesity (obese women), which is an important public health problem all over the world.

DETAILED DESCRIPTION:
Obesity is an important public health problem worldwide and is associated with non-communicable diseases such as Type 2 Diabetes, hypertension, coronary heart disease, hyperlipidemia, non-alcoholic fatty liver, some neoplasms, and infertility disease.However, it is supported by the literature that nutrition and obesity cause microbial dysbiosis.

In this study, it was aimed to use probiotics and yogurt with the thought that nutrition can manipulate the microbiota.

It was aimed to investigate the effects of probiotic yogurt consumption on anthropometric measurements, metabolic parameters, and gastrointestinal symptoms in obese women (25-45 years old) with the prospective method.

The study was carried out in patients who were diagnosed with obesity by the doctor, consulted the Dietitian, and accepted + signed the voluntary consent form.

Total data and measurements were followed and recorded by the same Dietitian. Compliance with medical nutrition therapy, recording of scales were followed weekly.Patients diagnosed with COVID-19 during the study were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 25-45 years, with a BMI of 27-35 kg/m2 diagnosed as obese by the doctor
* Female patients without a chronic disease
* Female patients between the ages of 25-45 with regular menstrual cycles,
* Female patients between the ages of 25-45 who are not pregnant or lactating
* Female patients who do not use drugs, herbal products, etc. nutritional supplements.

Exclusion Criteria:

* Patients with BMI≥ 36 kg/m2
* Patients with diabetes, gastrointestinal diseases, CRF, etc.
* Women in pregnancy and lactation period,
* Male patients
* Weight loss medicine etc. patients with drug use
* Patients who use antibiotics
* Patients using probiotics, propolis, herbal products, etc.
* Patients with menstrual irregularity
* Female patients who have entered the menopause

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The female gender was preferred in terms of ensuring homogeneity and sustainability of the diet.
Study Population: She was diagnosed with obesity by a doctor at Malatya Turgut Özal University Training and Research Hospital and was consulted to the Diet Polyclinic for appropriate Medical Nutrition Therapy; patients aged 25-45, female, with a BMI of 27 -35 kg/m2, who read and signed the voluntary consent form.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Determining Change in Obesity | 1 time per week/5 weeks
  * Mean percent change in initial and final body weight (kilogram)
  * Mean percent change initial and final waist circumference (cm):
  * Mean percent change initial and final waist/height ratio: It will be calculated by dividing waist circumference by height. The cut-off point of ratio will be taken as 0.5.
  * Mean percent change initial and final waist/hip ratio:The cut-off point for the Waist/Hip ratio, which was determined by dividing the waist circumference by the hip circumference, was determined as ≥0.90 cm for men and ≥0.85 cm for women.
  * Mean percent change initial and final fat mass: It measurement of individuals will be measured with the Body Composition Analyzer (in % and kg units). It is based on the difference in electrical permeability of fat-free tissue mass and fat.
  * Biochemical parameters was determined in mg/dL following the protocols established for: high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides and fasting glucose.

SECONDARY OUTCOMES:
Changes on the Gastrointestinal System | 1 time per week/5 weeks
  * Evaluation of the difference between individuals according to the Bristol Stool Scale. The Bristol Stool Scale is used to determine stool. The scale has seven stool types for visual identification of stool.
  * Gastrointestinal Symptom Rating Scale:The scale, which consists of 15 questions, includes questions about abdominal pain, heartburn, reflux nausea, dyspepsia and stool consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Sevan ÇETİN ÖZBEK, Study Director — Yüksek Ihtisas University
Locations (1):
- Malatya Training and Research Hospital, Malatya, Turkey (Türkiye)

REFERENCES:
- [Background] Cancello R, Turroni S, Rampelli S, Cattaldo S, Candela M, Cattani L, Mai S, Vietti R, Scacchi M, Brigidi P, Invitti C. Effect of Short-Term Dietary Intervention and Probiotic Mix Supplementation on the Gut Microbiota of Elderly Obese Women. Nutrients. 2019 Dec 10;11(12):3011. doi: 10.3390/nu11123011. PMID 31835452
- [Background] Wang ZB, Xin SS, Ding LN, Ding WY, Hou YL, Liu CQ, Zhang XD. The Potential Role of Probiotics in Controlling Overweight/Obesity and Associated Metabolic Parameters in Adults: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2019 Apr 15;2019:3862971. doi: 10.1155/2019/3862971. eCollection 2019. PMID 31118956
- [Background] Mazloom K, Siddiqi I, Covasa M. Probiotics: How Effective Are They in the Fight against Obesity? Nutrients. 2019 Jan 24;11(2):258. doi: 10.3390/nu11020258. PMID 30678355